CLINICAL TRIAL: NCT06795490
Title: Families in Balance: Enhancing Household Routines and Reducing Early Childhood Obesity Among Families With Low-income
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Bauer, Associate Professor of Nutritional Sciences, School of Public Health, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00263046; 1-R40-MC-53074-01-00 (Other Grant/Funding Number: Department of-Health Resources and Services Administration)
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Health Behavior
Keywords: Online program; Informational material; Surveys; Eating activity; Sleep; Health behaviors; Body mass index
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: About 150 adults and 150 children will take part in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Program (Experimental): Parents will participate in an online program.
  Interventions: Behavioral: Online program
- Control condition - Informational materials via email (Active Comparator): Parents will receive information via email.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Online program — Families in Balance Online is a 6-week online program that includes 6 weekly group discussions and 3 individual support sessions, all held over Zoom. Program activities will focus on improving parent and child self-regulation as a means to encourage healthy family mealtime, sleep, and screentime routines. Participants will engage in in person and online data collection activities to understand whether the program is impactful.
  Arms: Online Program
Behavioral: Control Condition — Families in Balance is an asynchronous program in which participants will be sent materials weekly over 6 weeks to encourage healthy family mealtime, sleep, and screentime routines. Participants will engage in in person and online data collection activities to understand whether the program is impactful.
  Arms: Control condition - Informational materials via email

SUMMARY:
This study will evaluate the effects of two different approaches to support healthy family mealtime, sleep, and screentime routines: A parent leader-guided online program that promotes parent and child self-regulation as a means to improve healthy family routines versus an asynchronous program that provides parents information about healthy family routines. Families will be randomly assigned to either of these programs and changes in parent and child outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Parents must be the legal and custodial guardian of a 2 through 5-year-old child
* Parents must report that their child is eligible for public health insurance
* Parents must be able to complete the study activities in English
* Parents must be able to complete study activities at a study location or at home, and online/via Zoom.

Exclusion Criteria:

- Children must not have serious medical problems that affect weight, sleep, activity, or eating.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Child age and sex-adjusted Body Mass Index (BMI) | Base line (pre-intervention) and approximately 5 months
  Differences in age- and sex-adjusted body mass index (BMI) among children of parents randomized to Families in Balance Online compared to children of parents randomized to Families in Balance at follow-up. Children's weight and height will be used to calculate BMI and measured using standardized protocols at baseline and follow-up.

SECONDARY OUTCOMES:
Child sleep duration | Base line (pre-intervention) and approximately 5 months
  This will be reported in minutes using data from surveys completed by parents.
Child daily screentime | Base line (pre-intervention) and approximately 5 months
  This will be reported in minutes using data from surveys completed by parents.
Child intake of key food groups | Base line (pre-intervention) and approximately 5 months
  This will be measured using a parent-completed 25-item dietary screener assessing intake of key foods/food groups (e.g., fruits and vegetables, sugar-sweetened beverages)
Child sleep routines | Base line (pre-intervention) and approximately 5 months
  This will be measured through parent completion of the Child Sleep Hygiene Scale which assesses 6 aspects of children's sleep/bedtime routines.
Child screentime limits | Base line (pre-intervention) and approximately 5 months
  This will be measured through parent completion of survey items measuring parents' limit setting with respect to screentime.
Family meal frequency | Base line (pre-intervention) and approximately 5 months
  This will be measured through parents' completion of survey items assessing the frequency with which families ate meals together.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bauer, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No